CLINICAL TRIAL: NCT01898910
Title: Ganglionated Plexi Ablation vs Renal Denervation in Patients Undergoing Pulmonary Vein Isolation. A Randomized Comparison
Brief Title: Ganglionated Plexi Ablation vs Renal Denervation in Patients Undergoing Pulmonary Vein Isolation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDGP-031
Record Dates: First submitted 2013-07-04; First posted 2013-07-15 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI+renal denervation+OMT (Active Comparator)
  Interventions: Procedure: PVI+renal denervation; Drug: Optimal medial therapy (OMT)
- PVI+GP ablation+OMT (Active Comparator)
  Interventions: Procedure: PVI + GP ablation; Drug: Optimal medial therapy (OMT)

INTERVENTIONS:
Procedure: PVI+renal denervation — After AF ablation procedure, the angiogram of both renal arteries is performed via femoral access. After that the treatment catheter is introduced into each renal artery and is applied discrete, radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm. After the procedure the control arterial angiogram should be done.
  Arms: PVI+renal denervation+OMT
Procedure: PVI + GP ablation — To accomplish ganglionated plexi ablation, LA target sites were identified as the anatomic locations where vagal reflexes were evoked by transcatheter high-frequency stimulation (HFS). Rectangular electrical stimuli were delivered at a frequency of 20-50 Hz, output amplitude 15 V and pulse duration of 10 ms, for 5 sec (Stimulator B-53, Biotok Inc, Russia).
  Arms: PVI+GP ablation+OMT
Drug: Optimal medial therapy (OMT) — Antiarrhythmic and antihypertensive therapy will be administered according to the guidelines

SUMMARY:
The investigators have conducted a prospective, double-blind, randomized study to assess the comparative safety and efficacy of two different strategies, PVI plus Renal Denervation (RD) versus PVI plus GP ablation, in patients with atrial fibrillation. Results were assessed after follow-up of at least 1 year with the use of an implanted monitoring device (IMD).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic drug-refractory AF (with history of failure of ≥ 2 class I or III antiarrhythmic drugs) in patients referred for catheter ablation of AF
* PAF with ≥1 monthly episodes or PersAF in patients who had already undergone ≥3 electrical cardioversions. PAF was defined as episodes lasting less than 7 days with spontaneous termination. PersAF was defined as lasting more than 7 days before being terminated pharmacologically or by electrical cardioversion.
* History of significant hypertension (defined as SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg), receiving treatment with at least one antihypertensive medication
* A glomerular filtration rate ≥45 mL/min/1⋅73 m2, with modification of diet using a renal disease formula

Exclusion Criteria:

* Previous atrial fibrillation ablation
* Type 1 of diabetes mellitus
* Structural heart disease
* Secondary cause of atrial hypertension
* Severe renal artery stenosis or renal arteries abnormalities
* Previous operations on renal arteries
* Pregnancy
* Previous heart, kidney, liver, or lung transplantation
* Unwillingness of participant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Freedom of AF or other atrial arrhythmias | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru